CLINICAL TRIAL: NCT04620343
Title: Exercise Induced Laryngeal Obstruction; a Randomized Controlled Treatment Trial
Brief Title: HelpILO - RCT on EILO Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/134444
Record Dates: First submitted 2020-10-09; First posted 2020-11-09 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Exercise Induced Laryngeal Obstruction (EILO)
Keywords: Larynx; Obstruction; Exercise
MeSH Terms: conditions — Laryngeal Diseases; Bites and Stings; Motor Activity | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Phase 1, Group 1 (Active Comparator): Patients are provided with basic information and breathing advice with biofeedback (IBA).
  This is the reference treatment against which the other methods will be measured.
  Interventions: Procedure: A: Breathing advice with bio-feedback
- Phase 1, Group 2 (Experimental): Patients are provided with basic information and breathing advice with biofeedback (IBA) and treated with inspiratory muscle training (IMT)
  Interventions: Procedure: B: Breathing advice with bio-feedback, Inspiratory muscle training (IMT)
- Phase 1, Group 3 (Experimental): Patients are provided with basic information and breathing advice with biofeedback (IBA) and treated with speech therapy
  Interventions: Procedure: C: Breathing advice with bio-feedback, Speech Therapy
- Phase 1, Group 4 (Experimental): Patients are provided with basic information and breathing advice with biofeedback (IBA) and treated with inspiratory muscle training (IMT) and speech therapy
  Interventions: Procedure: D: Breathing advice with bio-feedback, IMT and Speech Therapy
- Phase 2, Group 1 (No Intervention): Groups 2,3,4 in Phase 1 Wait for therapy effect
- Phase 2, Group 2 (Experimental): If patients from Phase 1, Group 1 (reference treatment) have unchanged CLE-scoring, they are treated with inspiratory muscle training (IMT) and speech therapy.
  Interventions: Procedure: A: If CLE-test unchanged, additional IMT and Speech Therapy
- Phase 3, Group 1 (Experimental): Treated with Surgery, supraglottoplasty - full procedure
  Interventions: Procedure: Surgery 1: Supraglottoplasty - full procedure under general anesthesia
- Phase 3, Group 2 (Experimental): Treated with Surgery, supraglottoplasty mini-invasive procedure
  Interventions: Procedure: Surgery 2: Supraglottoplasty - mini-invasive procedure under general anesthesia
- Phase3, Group 3 (No Intervention): Non-surgery control group

INTERVENTIONS:
Procedure: A: Breathing advice with bio-feedback — Information and breathing advice with biofeedback will serve as an active comparator in this study, and time allowed for IBA and biofeedback in this study will be max 30 min. The teaching will be provided by the attending physician and the test leader. The session will follow a strict checklist. After the laryngoscope has been secured in correct position the patient will be shown his/her larynx on the screen, providing the patient with basic knowledge on laryngeal anatomy and function in a calm atmosphere before the CLE-test. After, the patients will be trained to make any symptoms abate, and a good breathing posture and how to optimally use their breathing muscles.
  Arms: Phase 1, Group 1
Procedure: B: Breathing advice with bio-feedback, Inspiratory muscle training (IMT) — Breathing advise and IMT. The inspiratory muscle training (IMT) will build on the information the patients have obtained during the IBA and biofeedback session. The IMT will focus on training endurance and coordination of the PCA muscle, aiming to reduce fatigue of the abducting capacity of the larynx and to enhance coordination and create a sense of laryngeal control. When performing the IMT sessions, it is of utmost importance that a functional diaphragmatic breathing pattern has been established, and that this breathing pattern is maintained throughout all the IMT sessions. Once the patient has demonstrated that he/she is able to perform breathing according to these principles, the IMT session will follow a detailed protocol while wearing a flexible laryngoscope and settings and techniques are adjusted to ensure max open larynx. The patient will perform IMT training at home as instructed and have video meetings one and three weeks after initial training to observe progress.
  Arms: Phase 1, Group 2
Procedure: C: Breathing advice with bio-feedback, Speech Therapy — The training period with the speech therapist takes three days, divided into 6 sessions. The training is continued at home, implementing the techniques during physical activity and at rest. The aim of the speech therapy is to help the patients to develop a strategy on how to control his/her larynx during exercise, and to be able to continue exercising without experiencing dramatic EILO incidents. They will be informed that the best approach is to start practicing while performing low to moderate intensity exercise, and then gradually increase the intensity as they become more confident. It will be emphasized that the new breathing technique they are about to adopt will need to be repeated until it becomes adapted as a part of their automated breathing pattern. Patients will be followed up with video meetings one and three weeks after initial training to observe progress.
  Arms: Phase 1, Group 3
Procedure: D: Breathing advice with bio-feedback, IMT and Speech Therapy — All treatments as described above.
  Arms: Phase 1, Group 4
Procedure: A: If CLE-test unchanged, additional IMT and Speech Therapy — All treatments as described above.
  Arms: Phase 2, Group 2
Procedure: Surgery 1: Supraglottoplasty - full procedure under general anesthesia — Endoscopic supraglottoplasty with carbon dioxide laser and cold steel microlaryngeal instruments. The patient is intubated with an armored laser-tube which is positioned in the posterior midline to protect this area from laser injury. The laryngoscope is positioned into the vallecula and the surgery is visualized through an operation-microscope. CO2-laser beams of 2-4W focused with micro spot is utilized. Releasing incisions are made at the anterior border of both AEFs. The depth of the incisions are limited to the cranial border of the ventricular folds. The cuneiform tubercles including their surrounding mucosa are removed in a circular pattern before the two incisions are adjoined, thus creating a drop shaped excision. Care is taken to avoid scarring. It is recommended to protect the posterior commissure and the piriform sinus with wet tissue cloths. In case of perioperative edema of the laryngeal mucosa, corticosteroids are administrated to prevent laryngeal edema post-operatively.
  Arms: Phase 3, Group 1
Procedure: Surgery 2: Supraglottoplasty - mini-invasive procedure under general anesthesia — Endoscopic supraglottoplasty with carbon dioxide laser. The patients are intubated with an armored laser-tube, which is positioned in the posterior midline to protect this area from laser injury. The laryngoscope (Benjamin/Lindholm) is positioned into the vallecula and the surgery is visualized through an operation-microscope. CO2-laser beams of 2-4W focused with micro spot are utilized. Four punctures will be made along the lateral borders of both aryepiglottic folds bilateral, thus creating a row of small punctures parallel to the rim of the aryepiglottic folds. The punctions should not be deeper than the incision in the "full procedure" (above); i.e. less than 5 millimeter, and care must be taken to avoid heat affecting the nervus recurrens posteriorly. Care is taken to avoid scarring and collateral thermal injury. It is recommended to protect the posterior commissure and the piriform sinus with wet tissue cloths. No antibiotic prophylaxis is administered.
  Arms: Phase 3, Group 2

SUMMARY:
Exercise induced laryngeal obstruction (EILO) is a common cause of exertional breathing problems in young individuals, caused by paradoxical inspiratory adduction of laryngeal structures, and diagnosed by continuous visualization of the larynx during high intensity exercise.

DETAILED DESCRIPTION:
Exercise induced laryngeal obstruction (EILO) is a common cause of exertional breathing problems in young individuals, caused by paradoxical inspiratory adduction of laryngeal structures, and diagnosed by continuous visualization of the larynx during high intensity exercise.

Studies indicate that EILO responds positively to treatment interventions; however, the investigators lack randomized controlled studies to confirm this (10-15). This study aims to provide evidence-based information on interventions commonly applied to treat EILO. Background: Exercise induced laryngeal obstruction (EILO) is a common cause of exertional breathing problems in young individuals, caused by paradoxical inspiratory adduction of laryngeal structures, and diagnosed by continuous visualization of the larynx during high intensity exercise. Empirical data suggest that EILO consists of different subtypes that require different therapeutic approaches. However, currently applied treatment schemes do not rest on randomized controlled trials. This study aims to provide evidence-based information on treatment schemes commonly applied in patients with EILO.

Methods: Consenting patients consecutively diagnosed with EILO at Haukeland University Hospital will be randomized into four different conservative treatment arms, selected on the basis of promising reports from non-randomized studies: (A) standardized information and breathing advice only (IBA), (B) IBA plus inspiratory muscle training, (C) IBA plus speech therapy, and (D) IBA plus provision of both inspiratory muscle training and speech therapy. Differential effects in predefined EILO subtypes will be addressed. Patients failing the conservative approach and otherwise qualifying for surgical treatment by current department policy will be considered for randomization into (E) standard or (F) minimal laser supraglottoplasty, and a "wait-and-see" control group. Power calculations will be based on the main outcomes, laryngeal adduction during peak exercise, rated by a validated scoring system before and after the interventions.

Discussion: The study will provide evidence-based information on the treatment of EILO, listed as a priority in a recent statement issued by the European Respiratory Society, requested by clinicians and researchers engaged in this area, and relevant to 5-7% of young people.

ELIGIBILITY:
Inclusion Criteria:

* EILO with CLE score at peak exercise graded as ≥ 2 at glottic or supraglottic level and
* Respiratory complaints to an extent that the patient wants further treatment and follow-up.

Exclusion Criteria:

* Breathing problems caused by disorders other than EILO or well controlled asthma.
* Perceived to be unable to perform repeated maximal cardiopulmonary treadmill exercise tests, or failing to accept the procedures required for repeated successful CLE tests, or unable to perform any of the other examinations required by the protocol.
* Abnormal anatomy at rest in the laryngeal region or the upper airways.
* Age below 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaires | Day 1
  All patients will complete custom-made questionnaires recording demographic background variables and symptom scores. The questionnaires focus mainly on respiratory symptoms experienced by the patients, treatment they have been exposed to, and diagnoses they have been assigned. Relevant co-morbidities will also be recorded.
Pulmonary function and exercise test - Spirometry 1 | Through study completion, on average 6 months
  Recording of expiratory and inspiratory volumes and flows will be recorded: Forced expiratory and inspiratory volume capacity (FVC and FIVC). Volumes measured in liters
Pulmonary function and exercise test - Spirometry 2 | Through study completion, on average 6 months
  Recording of expiratory and inspiratory volumes and flows will be recorded: forced expiratory and inspiratory volume in first second (FEV1 and FIV1). Volumes measured in liters
Pulmonary function and exercise test - Spirometry 3 | Through study completion, on average 6 months
  Recording of expiratory and inspiratory volumes and flows will be recorded: forced expiratory and inspiratory flow at 50% of FVC (FEF and FIF50) and at 25-75% of FVC (FEF and FIF25-75). Volumes measured in liters.
Continuous Laryngoscopy Exercise test (CLE-test) and scoring | Through study completion, on average 6 months
  CLE-scores from the video recordings from the CLE-test will be evaluated. Two highly experienced raters will score all CLE tests according to a system that has been published previously. CLE scoring of glottic and supraglottic obstruction, grades 0 to 4.
Cardiopulmonary exercise (CPX) data - Variables of gas exchange | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Variables of gas exchange are measured breath-by-breath. Oxygen absorption measured in mL(min)/kg. Co2 production and O2 production in mL/min.
Cardiopulmonary exercise (CPX) data - duration of run | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Duration of run is recorded in minutes and seconds.
Cardiopulmonary exercise (CPX) data - distance of run | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Distance of run is recorded in meters
Cardiopulmonary exercise (CPX) data - oxygen consumption | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Variables of oxygen consumption will be recorded. Oxygen consumption is measured in (mL/min)/kg
Cardiopulmonary exercise (CPX) data - CO2 production | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Variables of CO2 production will be recorded in mL/minute.
Cardiopulmonary exercise (CPX) data - respiratory rates. | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Variables of respiratory and tidal volumes will be recorded in liters and ratios calculated.
Cardiopulmonary exercise (CPX) data - heart rates. | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Variables of heart rates will be recorded in Hf/min.
Cardiopulmonary exercise (CPX) data - Exercise tidal flow/volume loops | Through study completion, on average 6 months
  A treadmill will run according to a modified Bruce protocol, incrementing speed and/or grade every 1 min, aiming for peak oxygen uptake after 6-14 min. Exercise tidal flow/volume loops will be obtained at fixed interval during the session by plotting air flow (l/sec) and air volume the patient breathes during testing.
Continuous laryngoscopy exercise (CLE) with pressure recordings | During Phase 3, average duration 6 months.
  Translaryngeal resistance will be measured during CLE-testing in the third phase. Calculation of resistance will be based on pressure recordings obtained by two pressure sensors placed above and below the larynx, and airflow measured breath by breath by the mouth. Pressure is measured in kPa.

CONTACTS AND LOCATIONS:
Overall Officials: Hege H Clemm, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Children and Youth Clinic, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halvorsen T, Clemm HSH, Vollsaeter M, Roksund OD. Conundrums of Exercise-related Breathing Problems. Epiglottic, Laryngeal, or Bronchial Obstruction? Am J Respir Crit Care Med. 2020 Nov 15;202(10):e142-e143. doi: 10.1164/rccm.201910-1921IM. No abstract available. PMID 32783778
- [Background] Engan M, Engeseth MS, Fevang S, Vollsaeter M, Eide GE, Roksund OD, Halvorsen T, Clemm H. Predicting physical activity in a national cohort of children born extremely preterm. Early Hum Dev. 2020 Jun;145:105037. doi: 10.1016/j.earlhumdev.2020.105037. Epub 2020 Apr 11. PMID 32438296
- [Background] Fretheim-Kelly ZL, Halvorsen T, Clemm H, Roksund O, Heimdal JH, Vollsaeter M, Fintl C, Strand E. Exercise Induced Laryngeal Obstruction in Humans and Equines. A Comparative Review. Front Physiol. 2019 Oct 30;10:1333. doi: 10.3389/fphys.2019.01333. eCollection 2019. PMID 31736771
- [Background] Sandnes A, Hilland M, Vollsaeter M, Andersen T, Engesaeter IO, Sandvik L, Heimdal JH, Halvorsen T, Eide GE, Roksund OD, Clemm HH. Severe Exercise-Induced Laryngeal Obstruction Treated With Supraglottoplasty. Front Surg. 2019 Jul 31;6:44. doi: 10.3389/fsurg.2019.00044. eCollection 2019. PMID 31417908
- [Background] Sandnes A, Andersen T, Clemm HH, Hilland M, Vollsaeter M, Heimdal JH, Eide GE, Halvorsen T, Roksund OD. Exercise-induced laryngeal obstruction in athletes treated with inspiratory muscle training. BMJ Open Sport Exerc Med. 2019 Jan 18;5(1):e000436. doi: 10.1136/bmjsem-2018-000436. eCollection 2019. PMID 30792880
- [Background] Fretheim-Kelly Z, Halvorsen T, Heimdal JH, Strand E, Vollsaeter M, Clemm H, Roksund O. Feasibility and tolerability of measuring translaryngeal pressure during exercise. Laryngoscope. 2019 Dec;129(12):2748-2753. doi: 10.1002/lary.27846. Epub 2019 Jan 30. PMID 30698834
- [Background] Andersen TM, Sandnes A, Fondenes O, Clemm H, Halvorsen T, Nilsen RM, Tysnes OB, Heimdal JH, Vollsaeter M, Roksund OD. Laryngoscopy Can Be a Valuable Tool for Unexpected Therapeutic Response in Noninvasive Respiratory Interventions. Respir Care. 2018 Nov;63(11):1459-1461. doi: 10.4187/respcare.06674. No abstract available. PMID 30389835
- [Background] Clemm HSH, Sandnes A, Vollsaeter M, Hilland M, Heimdal JH, Roksund OD, Halvorsen T. The Heterogeneity of Exercise-induced Laryngeal Obstruction. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1068-1069. doi: 10.1164/rccm.201708-1646IM. No abstract available. PMID 29390192
- [Background] Roksund OD, Heimdal JH, Clemm H, Vollsaeter M, Halvorsen T. Exercise inducible laryngeal obstruction: diagnostics and management. Paediatr Respir Rev. 2017 Jan;21:86-94. doi: 10.1016/j.prrv.2016.07.003. Epub 2016 Jul 18. PMID 27492717
- [Background] Heimdal JH, Roksund OD, Halvorsen T, Skadberg BT, Olofsson J. Continuous laryngoscopy exercise test: a method for visualizing laryngeal dysfunction during exercise. Laryngoscope. 2006 Jan;116(1):52-7. doi: 10.1097/01.mlg.0000184528.16229.ba. PMID 16481809
- [Background] Maat RC, Roksund OD, Olofsson J, Halvorsen T, Skadberg BT, Heimdal JH. Surgical treatment of exercise-induced laryngeal dysfunction. Eur Arch Otorhinolaryngol. 2007 Apr;264(4):401-7. doi: 10.1007/s00405-006-0216-6. Epub 2007 Jan 4. PMID 17203312
- [Background] Maat RC, Roksund OD, Halvorsen T, Skadberg BT, Olofsson J, Ellingsen TA, Aarstad HJ, Heimdal JH. Audiovisual assessment of exercise-induced laryngeal obstruction: reliability and validity of observations. Eur Arch Otorhinolaryngol. 2009 Dec;266(12):1929-36. doi: 10.1007/s00405-009-1030-8. Epub 2009 Jul 8. PMID 19585139
- [Background] Roksund OD, Maat RC, Heimdal JH, Olofsson J, Skadberg BT, Halvorsen T. Exercise induced dyspnea in the young. Larynx as the bottleneck of the airways. Respir Med. 2009 Dec;103(12):1911-8. doi: 10.1016/j.rmed.2009.05.024. Epub 2009 Sep 26. PMID 19782550
- [Background] Maat RC, Hilland M, Roksund OD, Halvorsen T, Olofsson J, Aarstad HJ, Heimdal JH. Exercise-induced laryngeal obstruction: natural history and effect of surgical treatment. Eur Arch Otorhinolaryngol. 2011 Oct;268(10):1485-92. doi: 10.1007/s00405-011-1656-1. Epub 2011 Jun 5. PMID 21643933
- [Background] Sandnes A, Andersen T, Hilland M, Ellingsen TA, Halvorsen T, Heimdal JH, Roksund OD. Laryngeal movements during inspiratory muscle training in healthy subjects. J Voice. 2013 Jul;27(4):448-53. doi: 10.1016/j.jvoice.2013.02.010. Epub 2013 May 15. PMID 23683807
- [Background] Roksund OD, Heimdal JH, Olofsson J, Maat RC, Halvorsen T. Larynx during exercise: the unexplored bottleneck of the airways. Eur Arch Otorhinolaryngol. 2015 Sep;272(9):2101-9. doi: 10.1007/s00405-014-3159-3. Epub 2014 Jul 18. PMID 25033930
- [Background] Christensen PM, Heimdal JH, Christopher KL, Bucca C, Cantarella G, Friedrich G, Halvorsen T, Herth F, Jung H, Morris MJ, Remacle M, Rasmussen N, Wilson JA; ERS/ELS/ACCP Task Force on Inducible Laryngeal Obstructions. ERS/ELS/ACCP 2013 international consensus conference nomenclature on inducible laryngeal obstructions. Eur Respir Rev. 2015 Sep;24(137):445-50. doi: 10.1183/16000617.00006513. PMID 26324806
- [Background] Norlander K, Christensen PM, Maat RC, Halvorsen T, Heimdal JH, Moren S, Rasmussen N, Nordang L. Comparison between two assessment methods for exercise-induced laryngeal obstructions. Eur Arch Otorhinolaryngol. 2016 Feb;273(2):425-30. doi: 10.1007/s00405-015-3758-7. Epub 2015 Sep 8. PMID 26351037
- [Background] Hilland M, Roksund OD, Sandvik L, Haaland O, Aarstad HJ, Halvorsen T, Heimdal JH. Congenital laryngomalacia is related to exercise-induced laryngeal obstruction in adolescence. Arch Dis Child. 2016 May;101(5):443-8. doi: 10.1136/archdischild-2015-308450. Epub 2016 Feb 23. PMID 26906070
- [Background] Roksund OD, Olin JT, Halvorsen T. Working Towards a Common Transatlantic Approach for Evaluation of Exercise-Induced Laryngeal Obstruction. Immunol Allergy Clin North Am. 2018 May;38(2):281-292. doi: 10.1016/j.iac.2018.01.002. Epub 2018 Feb 19. PMID 29631736